CLINICAL TRIAL: NCT01983839
Title: Moxifloxacin Pharmacokinetic Profile and Efficacy Evaluation in the Empiric Treatment of Community-Acquired Pneumonia
Brief Title: PK Analysis of Moxifloxacin in the Treatment of CAP
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Kristina Öbrink-Hansen, MD, University of Aarhus
Other Study IDs: MOXI-274-13; 2007-58-0010 (Other: Datatilsynet, Denmark)
Record Dates: First submitted 2013-07-10; First posted 2013-11-14 (Estimated); Results first posted 2015-04-06 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-03

CONDITIONS: Pneumonia
Keywords: Moxifloxacin; Pneumonia; Pharmacokinetics
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pharmacokinetics Moxifloxacin: Patients with community-acquired pneumonia treated with moxifloxacin

SUMMARY:
At the Department of Infectious Diseases, Aarhus Denmark, moxifloxacin is used in the empirical treatment of severe community-acquired pneumonia (CAP). This study was designed to determine the pharmacokinetics of moxifloxacin 400 mg/day to patients treated empirically for CAP. To accomplish this aim, we established a pharmacokinetic population model. This approach was adopted with the dual purpose of assessing the potential efficacy of the drug and performing Monte-Carlo simulations to characterize the maximal MICs for which recommended pharmacokinetic-pharmacodynamic (PK-PD) targets are obtained for pathogens commonly known to cause CAP.

DETAILED DESCRIPTION:
We determined the pharmacokinetic profile of moxifloxacin 400 mg/day in 18 patients treated empirically for community-acquired pneumonia. . Moxifloxacin plasma concentrations were determined the day after therapy initiation using ultra high performance liquid chromatography. The moxifloxacin plasma concentration-time profiles were described with a one compartment model, using NONMEM. Peak drug concentrations (Cmax) and 24-hour area under the free drug concentration-time curve values (fAUC0-24) predicted for each patient were evaluated against epidemiological cut-off MIC values for Streptococcus pneumoniae, Haemophilus influenzae and Legionella pneumophilia. PK-PD targets adopted were Cmax/MIC ≥ 12.2 for all pathogens, fAUC0-24/MIC > 34 for S. pneumoniae and fAUC0-24/MIC > 75 for H. influenzae and L. pneumophilia. The same PK-PD estimates were used in the simulations of probability of target attainment (PTA) versus MIC.

ELIGIBILITY:
Inclusion Criteria:

* Patients with community-acquired pneumonia, treated with moxifloxacin

Exclusion Criteria:

* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with community-acquired pneumonia, treated with moxifloxacin, admitted to the Department of Infectious diseases, Aarhus University Hospital, Denmark
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2013-04; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eskild Petersen, MD, Assoc. Prof., D.Sc., Study Director — Department of Infectious Diseases, Aarhus University Hospital, Denmark
Locations (1):
- Department of Infectious Diseases, Aarhus University Hospital, Aarhus, Aarhus N, Denmark

REFERENCES:
- [Derived] Obrink-Hansen K, Hardlei TF, Brock B, Jensen-Fangel S, Kragh Thomsen M, Petersen E, Kreilgaard M. Moxifloxacin pharmacokinetic profile and efficacy evaluation in empiric treatment of community-acquired pneumonia. Antimicrob Agents Chemother. 2015 Apr;59(4):2398-404. doi: 10.1128/AAC.04659-14. Epub 2015 Feb 9. PMID 25666151

RESULTS

PARTICIPANT FLOW:
Groups:
- Pharmacokinetics Moxifloxacin: Patients with diagnosed CAP who were prescribed moxifloxacin 400 mg qd (Avelox® 400 mg Bayer) empirically by the treating physician, according to national CAP treatment guideline, had plasma concentrations of moxifloxacin determined. Patients under 18 years of age were excluded from the study and the age, gender and body weight of each enrolled patient were registered.
Period: Overall Study
Arm/Group | Pharmacokinetics Moxifloxacin
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pharmacokinetics Moxifloxacin
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 14
  >=65 years | 3
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 73 [66 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 8
Body weight [Median (Inter-Quartile Range); unit: kg] | 72.6 [64.1 to 80.6]

OUTCOME MEASURES:

1. Primary Outcome: Total Peak Plasma Concentration (Cmax)
Description: The moxifloxacin plasma concentration-time profiles were described with a one compartment model with first-order absorption and elimination rate. The model estimated median values of total Cmax for the current study population were reported.
  Each individual model predicted Cmax were divided by the ECOFF MIC for S. pneumoniae (0.5 mg/L), H. influenzae (0.125 mg/L) and L. pneumophilia (1.0 mg/L)
Time Frame: The second day of Moxifloxacin treatment
Measure: Median (Inter-Quartile Range); unit: mg/L
Groups:
- Pharmacokinetics Moxifloxacin: Patients with diagnosed CAP who were prescribed moxifloxacin 400 mg qd (Avelox® 400 mg Bayer) empirically by the treating physician, according to national CAP treatment guideline, had plasma concentrations of moxifloxacin determined. Patients under 18 years of age were excluded from the study and the age, gender and body weight of each enrolled patient were registered.
  The model estimated median values of total Cmax and fAUC0-24 for the current study population were3.99 mg/L (IQR 3.19; 5.29) and 32.78 mg.hr/L (IQR 22.75; 47.31). respectively.
Arm/Group | Pharmacokinetics Moxifloxacin
Number analyzed (Participants) | 18
mg/L | 3.99 [3.18 to 5.29]

2. Primary Outcome: Area Under the Free Concentration-time Curve (fAUC0-24)
Description: The moxifloxacin plasma concentration-time profiles were described with a one compartment model with first-order absorption and elimination rate. The model estimated median values of fAUC0-24 for the current study population were reported.
  fAUC0-24 were divided by the ECOFF MIC for S. pneumoniae (0.5 mg/L), H. influenzae (0.125 mg/L) and L. pneumophilia (1.0 mg/L)
Time Frame: The second day of Moxifloxacin treatment
Population: The model estimated median values of fAUC0-24 for the current study population were32.78 mg.hr/L (IQR 22.75; 47.31). respectively.
Measure: Median (Inter-Quartile Range); unit: mg.hr/L
Arm/Group | Pharmacokinetics Moxifloxacin
Number analyzed (Participants) | 18
mg.hr/L | 32.78 [22.75 to 47.31]

ADVERSE EVENTS:
Description: Serious and non-serious adverse events were not collected.
Arm/Group | Pharmacokinetics Moxifloxacin
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes